CLINICAL TRIAL: NCT06344884
Title: Early Patient Removal of Urinary Catheters After Urogynecologic Surgery
Acronym: CARES2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-2619
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Urinary Retention Postoperative; Postoperative Urinary Tract Infection; Catheter Site Pain

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Catheter Removal (Experimental): Participants in this arm will be asked to remove their catheters POD1.
  Interventions: Procedure: Early catheter removal
- Standard Catheter Removal (No Intervention): Participants in this arm will be asked to remove their catheters POD3-4.

INTERVENTIONS:
Procedure: Early catheter removal — Catheter removal the day after surgery as opposed to standard of care (3 to 4 days after surgery)
  Arms: Early Catheter Removal

SUMMARY:
Management of postoperative urinary retention often requires the use of indwelling catheters. In a previous study, the investigators determined that patient removal of catheters at home is non-inferior to standard office removal on postoperative day three or four (POD3-4). The purpose of this study is to determine whether patient removal of catheters at home on postoperative day one (POD1) is noninferior to removal on POD 3-4.

DETAILED DESCRIPTION:
Randomized, controlled, non-inferiority trial to compare the risk of urinary retention between patient urinary catheter removal on POD1 versus POD3-4 after urogynecologic surgery.

Aim One: Is the risk of urinary retention non-inferior with patient removal of transurethral catheters on POD1 versus POD3-4 after urogynecologic surgery?

Aim Two: Does healthcare resource utilization (nursing calls, patient messages, and office visits) differ between patient removal of transurethral catheters on POD1 versus POD3-4?

Aim Three: Does the patient experience differ between patient removal of transurethral catheters on POD1 versus POD3-4?

Aim Four: Does the incidence of postoperative UTI differ between patient removal of transurethral catheters on POD1 versus POD3-4?

Aim Five: Does the risk of delayed or recurrent postoperative urinary retention differ between patient removal of transurethral catheters on POD1 versus POD3-4?

Screening: Preoperative clinics at UNC Rex Urogynecology will be screened for all women who are undergoing a prolapse or anti-incontinence procedure.

Study Treatment/Intervention

Postoperatively if patients fail their voiding trial in the post-anesthesia care unit (PACU) and are willing to perform home catheter removal after instruction

Patients will be randomized to a catheter management arm: self-catheter removal on POD1 or POD3-4

POD 1 - Patients in the intervention arm will be reminded to remove their catheters

They will be instructed to remove their urinary catheter at 0700 and to call the clinic office by noon if they have not voided

If they are unable to void or have any other concerning symptoms, they will be scheduled for a same day nurse visit

Patients who are unable to void will then be taught clean intermittent self-catheterization, per usual management of postoperative voiding dysfunction

POD 3 (or by POD 4 for Thursday cases) - Patients in the control arm will be reminded to remove their catheters

* Patients undergoing surgery on Thursday will perform catheter removal on Monday. This is what was done in previous studies in order to prevent resource over-utilization on weekends. Patients undergoing surgery on Wednesday (typically only rare add-on cases) will be excluded.

They will be instructed to remove their urinary catheter at 0700 and to call the clinic office by noon if they have not voided

If they are unable to void or have any other concerning symptoms, they will be scheduled for a same day nurse visit

Patients who are unable to void will then be taught clean intermittent self-catheterization, per usual management of postoperative voiding dysfunction

Week 2 Phone Call

Patients will be called by study personnel to check in on any voiding symptoms or issues and complete phone survey regarding the following categories: Pain, Ease of use, Satisfaction, Likelihood to use again.

Week 6 Visit

Patients will have a standard office visit around 6 weeks postoperatively. At this visit, a post-void residual assessment will be performed.

Follow-up through postoperative visit after surgery

Postoperative complications, such as urinary tract infection (UTI) or delayed urinary retention will be monitored from the chart

Patients will be randomized on the day of surgery. Each subject's participation will last from the day of surgery to the day of catheter removal (on POD 1-4). They will also be called two weeks postoperatively for a check-in and survey over the phone. Postoperative complications will be monitored until their postoperative visit at 6-8 weeks after surgery.

The recruitment and data collection period is expected to last one year. The entire study including data collection, analysis and publication will take up to 3 years. -

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing prolapse or anti-incontinence surgery who fail their voiding trials prior to discharge.

Exclusion Criteria:

* Non-English speaking (due to limited resources to consent non-English speaking patients)
* Pregnant
* Postvoid residual (PVR) >150 mL or dependent upon catheterization to void pre-operatively
* Intra-operative complication requiring prolonged catheterization

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Number of patients with ongoing urinary retention (noninferiority) | From Postoperative day 1 through postoperative week 8
  Defined as need for catheter replacement or clean intermittent self catheterization (CISC) after catheter removal on POD1 vs POD3-4. A 95% confidence interval of the difference in proportions between the two groups will be used to assess the tenability of a non-inferiority proposition.

SECONDARY OUTCOMES:
Number of patient contacts for voiding dysfunction by Type | From Postoperative day 1 through postoperative week 8
  Nursing calls, patient messages, and/or office visits will be summarized.
Total patient contacts for voiding dysfunction Combined | From Postoperative day 1 through postoperative week 8
  The total number of nursing calls, patient messages, and/or office visits combined.
Number of patients treated for postoperative UTI. | From Postoperative day 1 through postoperative week 8
  A case of postoperative UTI will be defined by patient receiving antibiotic treatment for UTI. This typically happens as a result of patient symptoms and/or a positive urine culture.
Number of patients with ongoing urinary retention | From Postoperative day 1 through postoperative week 8
  Defined as need for catheter replacement or clean intermittent self catheterization (CISC) after catheter removal on POD 1 vs 3-4.
Patient Satisfaction Survey Score-Pain | Postoperative week 2
  One survey question will be asked regarding Pain on a Likert Scale. The question is scored 0-4 with a higher score representing more pain.
Patient Satisfaction Survey Score-Ease of Use | Postoperative week 2
  One survey question will be asked regarding Ease of use on a Likert Scale. The question is scored 0-4 with a higher score meaning more difficulty or a worse outcome.
Patient Satisfaction Survey Score-Satisfaction | Postoperative week 2
  One survey question will be asked regarding Satisfaction on a Likert Scale. The question is scored 0-3 with a higher score meaning more satisfied or a better outcome.
Patient Satisfaction Survey Score-Likelihood to Use Again | Postoperative week 2
  One survey question will be asked regarding likelihood to use again on a Likert Scale. The question is scored 0-3 with a higher score meaning more likely or a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Tholemeier, MD, Principal Investigator — University of North Carollina at Chapel Hill
Locations (1):
- UNC Health Rex, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.